CLINICAL TRIAL: NCT01186224
Title: A Comparison of Plerixafor/G-CSF With Chemotherapy/G-CSF for Stem Cell Mobilisation
Brief Title: Plerixafor Harvesting And No Chemotherapy for Transplantation of Autologous STem Cells In Cancer (PHANTASTIC)
Acronym: PHANTASTIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Liverpool (Other)
Collaborators: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PHANTASTIC; 2009-013798-16 (EudraCT Number)
Record Dates: First submitted 2010-08-18; First posted 2010-08-23 (Estimated); Last update posted 2025-03-17 (Actual); Status verified 2010-02

CONDITIONS: Multiple Myeloma; Plasma Cell Dyscrasia; Lymphoma; Lymphoproliferative Disorders
MeSH Terms: conditions — Multiple Myeloma; Paraproteinemias; Lymphoma; Lymphoproliferative Disorders | interventions — plerixafor; Granulocyte Colony-Stimulating Factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Plerixafor plus G-CSF for patients undergoing stem cell harvesting (Experimental): Single arm comparison of plerixafor plus G-CSF for patients undergoing stem cell harvesting
  Interventions: Drug: Plerixafor and G-CSF

INTERVENTIONS:
Drug: Plerixafor and G-CSF — G-CSF will be given daily from day 1, which will usually be timed to fall toward the end of the working week. Plerixafor will commence on day 4 at as near to 10 PM as practicable, and also on day 5 and subsequent days (maximum of 4 total days) at a similar time of day if insufficient CD34+ cells have been collected. Stem cell harvesting will be carried out on day 5 and if necessary on days 6, 7 and 8, until the target yield of 4 x 106 CD34+ cells /kg recipient weight have been achieved.
  The daily dose of G-CSF is 300 ug for patients up to and including 60kg in weight; 480 ug for patients over 60 kg but under 96 kg, and 600 ug for patients weighing 96 kg or more. This equates to a dose of at least 5 ug/kg (maximum 8 mg/kg) for all patients up to 120 kg. The daily dose of plerixafor is 240 ug/kg if the creatinine clearance is equal to or greater than 50mls/minute; if less than this then the dose is 160 ug/kg daily.

SUMMARY:
To assess the efficacy and toxicity of plerixafor (AMD 3100) together with granulocyte-colony stimulating factor (G-CSF) for stem cell mobilisation, in patients with myeloma or lymphoma requiring high dose chemotherapy with stem cell rescue.

ELIGIBILITY:
Inclusion Criteria:

* All of the following must be satisfied:

Aged 18 or over

Able to give informed written consent.

Diagnosis of EITHER multiple myeloma or related plasma cell dyscrasia, OR any form of lymphoma or associated lymphoproliferative disease Autologous stem cell transplantation is planned as the next course of treatment.

The patient has not previously undergone a mobilisation attempt for the current transplant. Patients who have received previous autologous transplants at least 2 years previously are eligible, as long as stem cell mobilisation has not been attempted for the current transplant.

No serious concomitant illness (e.g. heart disease) that might preclude completion of the study.

Creatinine clearance of at least 30 mls/min. Note that a dose reduction of plerixafor is required where the creatinine clearance is between 30-50 mls/min; see section 3.3/5.1/5.3.

Negative pregnancy test in women of childbearing age.

Exclusion Criteria:

* Unable to give informed written consent

Pregnancy or lactating

Creatinine clearance of less than 30 mls/min. Patients with clearances lower than this may still be able to receive plerixafor at reduced dosage following discussion with the trial co-ordinators, but are not eligible for entry into this trial.

Any previous attempt at mobilisation for the current transplant. Patients with any form of leukaemia, INCLUDING PLASMA CELL LEUKAEMIA, are not eligible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2010-05 (Actual); Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
A composite primary endpoint of BOTH an adequate stem cell harvest (≥4 x 106 CD34+/kg in no more than 2 aphereses); AND a neutrophil count that never falls below 1.0 x 109 / Litre in the 3 weeks following initiation of mobilisation. | 3 weeks following initiation of mobilisation

SECONDARY OUTCOMES:
Serial neutrophil and platelet counts during mobilisation | 1 Day
Total stem cell yield in 1-2 aphereses | 1 day
The usage of plerixafor and the number and timing of apheresis collections | 1 day
The time to neutrophil engraftment after subsequent transplantation | First of 2 consecutive days on which the neutrophil count equals or exceeds 0.5 x 109/litre
The time to platelet engraftment after subsequent transplantation | First of two consecutive days on which the platelet count equals or exceeds 50 x 109/litre, having been free of platelet transfusion for at least 48 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Dept of Haematology, University of Liverpool, Liverpool, Merseyside, United Kingdom